CLINICAL TRIAL: NCT01834053
Title: Safety and Efficacy of Bone Marrow Derived MNCs for the Treatment of Huntingtons Chorea. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Safety and Efficacy of Bone Marrow Derived MNCs for Treatment of Cells for the Treatment of Hunting Tons Chorea.
Acronym: BMACHC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, CO-Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00106
Record Dates: First submitted 2013-04-11; First posted 2013-04-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Huntington Disease
Keywords: Huntington Disease,stem cell therapy
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STEM CELL (Other): Transfer of autologous Stem cell( MNCs) intrathecally
  Interventions: Biological: autologous Stem Cell

INTERVENTIONS:
Biological: autologous Stem Cell — Intrathecal transplantation of autologous 100 millions Stem cells{MNCs } per dose'
  Other Names: Intrathecal transplantation of autologous MNCs

SUMMARY:
This study is Single arm, Single Centre trial to check the Safety and Efficacy of Bone Marrow Derived Autologous mononuclear cell {MNC} (100 Million per dose).trial to be conducted for 36 months in patients with diabetes Mellitus in India,Primary outcome measure are Improvement in cognitive and Psychiatric Symptoms and Improvement in Jerky,random, and Uncontrollable Movements called Chorea.

DETAILED DESCRIPTION:
This study is Single arm, Single Centre trial study the Safety and Efficacy of Bone Marrow Derived Autologous mononuclear cells (MNCs) ,to be conducted for 36 months in patients with diabetes Mellitus in India,Primary outcome measure are Improvement in cognitive and Psychiatric Symptoms and Improvement in Jerky,random, and Uncontrollable Movements called Chorea.

ELIGIBILITY:
Inclusion Criteria:

* Patient should suffer from Hunting tons Chorea,
* Hunting tons chorea commonly become noticeable between the ages of 35 -44
* Willingness to undergo Bone Marrow derived Autologous cell Therapy.
* Ability to comprehend the explained protocol and thereafter give an informed consent as well as sign the required Informed Consent form(ICF) for the study.
* Ability and willingness to regular visit to hospital for protocol procedures and follow up

Exclusion Criteria:

* Patient with History of Immunodeficiency HIV+,Hepatitis B virus ( HBV) and History of Life threatening allergic or immune -Mediated Reaction. the site of bone marrow aspiration potentially limiting Procedure.
* alcohol and drug abuse / dependence.
* Severe skin infection.
* Haemodynamically unstable.

  =subject with primary and secondary diabetes , Insulin dependence.
* Neurological disease caused by autoimmune or genetic cause.
* patients suffering from peripheral muscular dystrophy.

Ages: 35 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in Cognitive and psychiatric symptoms | 6 Months

SECONDARY OUTCOMES:
Improvement in neuropsychiatric behaviour | 6 Months
Increase in life expectancy | 6 Months
  Increase in life expectancy.Time period- 6 Months
Improvement in writhing motions or abnormal posturing | 6 month
  -Improvement in writhing motions or abnormal posturing
Improvement in compulsive behaviour | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, M.S, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India